CLINICAL TRIAL: NCT00693641
Title: Efficiency of a Jellyfish Sting Inhibitor Sun Lotion and Protocols for Jellyfish Sting Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Chief Physician Kim Alexander Tønseth, Rikshospitalet HF
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-02-12-1 (UIO, BIOLOGEN); 2008-001519-39 (SLV)
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Pain
Keywords: Jellyfish; Cyanea sp; Safe Sea; Prevention; treatment; Pain relief; Prevention of pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Safe Sea™ jellyfish sting inhibitor (barrier, or "repellent") lotion
  Interventions: Other: Safe Sea sun lotion with jellyfish sting protection SPF 15
- 2 (Placebo Comparator): Regular sun lotion
  Interventions: Other: Nivea sun, caring sun lotion SPF 15

INTERVENTIONS:
Other: Safe Sea sun lotion with jellyfish sting protection SPF 15 — Prevent or significantly reduce jellyfish sting using sun lotion with a jellyfish sting inhibitor. The amount of lotion applied to the skin before spreading is the same as for regular sun lotion 2.00 mg.cm-²± 2.5%.
  Other Names: SunCare sunlotion with jellyfish sting protection SPF 15
  Arms: 1
Other: Nivea sun, caring sun lotion SPF 15 — The amount of lotion applied to the skin before spreading is 2.00 mg.cm-²± 2.5%.
  Arms: 2

SUMMARY:
The purpose of the study is to investigate the effectiveness of a sun lotion containing a specific Jellyfish sting inhibitor versus regular sun lotions as controls. In addition, to investigate the effectiveness of hot/cold immersion for the treatment of Cyanea sp stings versus local pain relief with prescription free pharmaceutical drug (Xylocain 30 mg/ml (3%) lidocain).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* men or women
* aged 18 or over

Exclusion Criteria:

* People with atopic diseases, e.g., asthma, allergic rhinorrhea or rhinitis, hay fever, or atopic skin inflammation
* People who suffer from skin diseases in the testing regions or whose inner forearms are too hairy to allow for interpretation of the test
* People who have used any medical or cosmetic product on either arm for 48 hours before the start of the experiment
* People who are taking antihistamines or steroids
* Subjects with medical conditions which, in the opinion of the investigator, pose risks that would prohibit participating
* Subjects with a history of keloid formation will be excluded from the Jellyfish protocol
* Subjects with allergy to lidocain or other local pain substances

If the arms contain hair that might reduce the jellyfish tentacle contact with the skin, the arm must be shaved in advance, so the skin has no sign of piling or any skin damage before the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The purpose of the study is to investigate the effectiveness of a sun lotion containing a specific Jellyfish sting inhibitor versus regular sun lotions or no protection at all when in contact with Cyanea SP. | Repeated jellyfish contact for total of 240 second or until pain occurs
  We want to find out how much longer it takes before you get stung if one at all gets stung when you have a protective layer on the skin. We also want to find out if the reduction in pain is significantly less when the skin has jellyfish protection using visual analog scale (VAS).

SECONDARY OUTCOMES:
Investigate the effectiveness of hot/cold immersion for the treatment of Cyanea sp stings versus local pain relief with prescription free pharmaceutical drugs called Xylocain with lidocaine | Pain relief treatment will start after 10 minutes, repeat treatment after 30 minutes if VAS score > 10.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Karlsen, Associate prof., Study Director — University of Oslo, Biologisk Stasjon Drøbak
Locations (1):
- University of Oslo, Biologisk Stasjon Drøbak, Biologveien 2, Drøbak, Norway